CLINICAL TRIAL: NCT01245075
Title: Deep Brain Stimulation of the Nucleus Accumbens as a Novel Treatment in Severe Opioid Addiction
Acronym: NASA
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jens Kuhn (Other)
Responsible Party: Sponsor-Investigator, Jens Kuhn, Prof. Dr., University of Cologne
Organization: University of Cologne (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10-090
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Addiction
MeSH Terms: conditions — Behavior, Addictive | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Brain Stimulation (Active Comparator): Stimulator setting is ON
  Interventions: Other: Deep brain stimulation
- Placebo (Sham Comparator): Stimulator setting is OFF
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Deep brain stimulation — Deep brain stimulation on
  Arms: Deep Brain Stimulation
Other: Placebo — deep brain stimulation off
  Arms: Placebo

SUMMARY:
The main objective of this study is to assess the efficacy of bilateral deep brain stimulation (DBS) of the Nucleus accumbens (NAc) as a novel treatment in severe opioid addiction. The included patients have been treated so far with a substitute in form of methadone.

Our hypothesis is that bilateral DBS of the NAc will significantly reduce the craving for heroin and thus enable the patients to decrease their Levomethadone-dosage substantially.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Proficiency in the German language
* Long lasting heroin addiction (fulfilled diagnostic-criteria according to DSM-IV,ICD-10)
* At least one detoxication-treatment without a long-term period of abstinence has already taken place
* Long-term inpatient treatment to support abstinence have occurred
* Free patient's decision / Informed Consent (existing comprehensive ability in meaning, methodology and execution of the study and ability of acceptance)
* If prior medication, stable dosage of psychopharmacological drugs over the last three months, which shall, after checking be retained during the study
* Substitution treatment with constant dose within the last three months before study inclusion

Exclusion Criteria:

* Hospitalization by PsychKG
* Clinical relevant psychiatric comorbidity (schizophrenic psychoses, bipolar affective diseases, severe personality disorder)
* Contraindications of a MRI-examination, e.g. implanted cardiac pacemaker/ heart defibrillator
* Current and in the last six months existent paranoid-hallucinated symptomatology
* Foreign aggressiveness in the last six months
* Verbal IQ < 85 (evaluated with the German Mehrfachauswahl-Intelligenz-Test (MWT-A/B))
* Stereotactic respectively neurosurgical intervention in the past
* Neoplastical neurological diseases
* Contraindications of a stereotactic operation, e.g. increased bleeding-disposition, cerebrovascular diseases (e.g. arteriovenous malfunction, aneurysms, systemic vascular diseases)
* Serious and instable organic diseases (e.g. instable coronal heart disease)
* tested positively for HIV
* pregnancy and/or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of Levomethadone | seven month
  Reduction of the dosage of the substitute (in detail Levomethadone) comparing baseline and the particular ward rounds during and at the end of the crossover-design.

SECONDARY OUTCOMES:
Drug seeking, goal directed behavior, Craving, Psychological components Laboratory parameters in the urine (parallel consumption of other drugs) | seven month
  Drug seeking and goal directed behavior (accessed with EEG) Craving (10-point visual analog scale (VAS)) Psychological components (Anxiety (HAMA); Depression (BDI-II); Quality of life (MSLQ) . Laboratory parameters in the urine (parallel consumption of other drugs)

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Visser-Vandewalle, MD, Principal Investigator — University of Cologne; Jens Kuhn, MD, Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, Cologne, Germany

REFERENCES:
- [Derived] Baldermann JC, Schuller T, Huys D, Becker I, Timmermann L, Jessen F, Visser-Vandewalle V, Kuhn J. Deep Brain Stimulation for Tourette-Syndrome: A Systematic Review and Meta-Analysis. Brain Stimul. 2016 Mar-Apr;9(2):296-304. doi: 10.1016/j.brs.2015.11.005. Epub 2015 Dec 29. PMID 26827109